CLINICAL TRIAL: NCT01884012
Title: Effect of Long-term Oxygen Therapy on Exercise Capacity and Quality of Life in Patients With Pulmonary Arterial and Chronic Thromboembolic Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEK 2012-0538
Record Dates: First submitted 2013-05-13; First posted 2013-06-21 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Arterial and Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplemental oxygen (Experimental): Supplemental oxygen 3 liters/minute given via a nasal cannula for 16 hours a day
  Interventions: Procedure: long term oxygen therapy
- Sham room air (Sham Comparator): Room air given at a flow rate of 3 liters per minute for 16 hours a day
  Interventions: Procedure: long term oxygen therapy

INTERVENTIONS:
Procedure: long term oxygen therapy

SUMMARY:
In this randomized-controlled, cross-over trial the investigators test the effect of long-term oxygen therapy (> 16h/day) given for 5 weeks with a wash-out period between phases of 2 weeks on exercise performance and quality of life and many physiological parameters in patients with pulmonary arterial and chronic thromboembolic pulmonary hypertension.

ELIGIBILITY:
Inclusion criteria:

- Adult patients with established diagnosis of pulmonary arterial or chronic thromboembolic pulmonary hypertension (class I and IV according to the latest WHO classification scheme of Dana Point 2008) on optimized medical therapy and in stable condition for at least 4 weeks, who desaturate in the 6 minute walking test by =4% to values <92%.

Exclusion criteria:

* Patients in unstable conditions requiring frequent therapeutic adaption
* pregnant women
* patients with pulmonary venous hypertension due to left heart diseases
* patients with relevant concomitant lung disease and severe daytime hypoxemia

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | 5 weeks
  6 minute walk distance according to american thoracic society (ATS) guidelines
Quality of life | 5 weeks
  QoL assessed by the short form of the medical outcome questionnaire (SF-36) physical functioning scale

SECONDARY OUTCOMES:
Daily activity | 5 week
  measured by actigraphy
hemodynamics by echocardiography | 5 weeks
  Full echocardiographic assessment
quality of life | 5 weeks
  SF-36
arterial blood gas | 5 weeks
  partial pressure of oxygen (PaO2)
operating hours of oxygen concentrator | 5 weeks
  efficacy of oxygen treatment
mean nocturnal oxygen saturation | 5 weeks
  Ambulatory Sleep Study
tests of cognitive performance | 5 weeks
  STROOP-Test
Quality of life | 5 weeks
  Minnesota living with heart failure questionnaire
Venous blood | 5 weeks
  N-terminal brain natriuretic peptide (NT-proBNP)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich Somaini, MD, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Canton of Zurich, Switzerland